CLINICAL TRIAL: NCT03108742
Title: Randomized Control Study of Dermal Staples vs Subcuticular Sutures on Postoperative Scar After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Dongsik Bae, Professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-12-010-001
Record Dates: First submitted 2017-03-20; First posted 2017-04-11 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Thyroidectomy; Pain; Esthetic; Dermal Stapler
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dermal stapler (Experimental)
  Interventions: Device: INSORB
- classic intradermal suture (Active Comparator)
  Interventions: Procedure: classic intradermal suture

INTERVENTIONS:
Device: INSORB — dermal stapler for skin closure
  Arms: dermal stapler
Procedure: classic intradermal suture — intradermal suture for skin closure
  Arms: classic intradermal suture

SUMMARY:
In this study, a randomized controlled study was conducted between two groups of 20 classic recipients of intradermal sutures and 20 recipients of intradermal staple methods for patients undergoing the same cervical incision. This is a study to see if there is any difference in pain and esthetics in scar formation of these groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient who will have thyroid surgery

Exclusion Criteria:

1. done thyroid surgery before
2. done any radiotherapy on neck
3. who needs neck dissection
4. laparoscopic ot robotic surgery
5. under 18 years old or over 70 years old
6. bad general condition, high American Society of Anesthesiologists (ASA) score (over 3)
7. who used immunosuppressive drugs in 6 months
8. breast feeder or pregnancy
9. who disagrees to do this trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Modified Stony Brook Scar Evaluation Scale (SBES) | Change from Baseline scar at 6 months
  Evaluate scar
Manchester Scar Scale (MSS) | Change from Baseline scar at 6 months
  Evaluate scar
Visual Analogue Scale (VAS) | Change from Baseline pain at 6 months
  Evaluate pain

CONTACTS AND LOCATIONS:
Locations (1):
- Dongsik Bae, Busan, South Korea